CLINICAL TRIAL: NCT02440438
Title: Factors Associated With Relapses in Patients Suffering From Clostridium Difficile Infection: Immune Response
Brief Title: Host Immune Response to Clostridium Difficile Infection (ICD)
Acronym: ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013.806
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Diarrhea Due to Clostridium Difficile
Keywords: Clostridium difficile, recurrence, relapse, antibodies, immune response, prognosis
MeSH Terms: conditions — Recurrence | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clostridium difficile infection (Experimental)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood samples of 10 mL will be performed every 2 days from the first symptoms of CDI and until clinical recovery and/or hospital discharge

SUMMARY:
Clostridium difficile is responsible for up to 25% of reported antibiotic associated diarrhea cases and virtually all cases of pseudomembranous colitis (PMC). The clinical spectrum of C. difficile infection (CDI) varies in severity from asymptomatic carriage to self-limited, mild, watery diarrhea, to PMC, intestinal perforation, toxic megacolon, sepsis, fulminant colitis, and death. In the past decade, the 027/NAP1/BI strain has emerged world-wide and has been implicated in large outbreaks with increased severity, frequent recurrence, and significant mortality. The host immune responses can influence the severity of CDI and play crucial roles in CDI onset, progression, and overall prognosis. Low serum concentrations of antibodies directed against the toxins A&B of C. difficile have been associated with a higher risk of recurrence. However, there are conflicting reports.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized
* Suffering from diarrhea related to C. difficile
* Confirmed diagnosis of CDI
* Informed consent by the patient
* Affiliated to the social security regime

Exclusion Criteria:

* Out-patient
* No confirmed diagnosis of CDI
* Decline of participation
* Patient not affiliated to the social security regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
immune response rate | up to 60 days after diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Hygiène, Epidémiologie et Prévention - Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] P Vanhems. "État des lieux des pratiques de prise en charge des ICD en France - Réseau DIFTEC" - JNI 2017 (symposium).
- [Result] "Incidence des infections à C. difficile" - communication (HCL Lyon, services d'Hygiène & Microbiologie). Auteurs indiqués : P. Vanhems, L. Oltra, M. Hulin, F. Vandenesch, O. Dauwalder.